CLINICAL TRIAL: NCT03672747
Title: The Impact of Spontaneous Cortical Activity on Neural Oscillations and Behavioral Performance: Evidence From High-definition tDCS and MEG
Brief Title: Modulation of Spontaneous Cortical Activity by tDCS: BRAIN Initiative I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 0580-18-FB; RF1MH117032 (NIH)
Record Dates: First submitted 2018-08-15; First posted 2018-09-14 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Brain Function
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Full crossover; all participants complete all conditions
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Anodal Brain Stimulation (Active Comparator): Participants will receive anodal stimulation using high-definition tDCS
  Interventions: Device: transcranial direct-current stimulation (tDCS)
- Cathodal Brain Stimulation (Active Comparator): Participants will receive cathodal stimulation using high-definition tDCS
  Interventions: Device: transcranial direct-current stimulation (tDCS)
- Sham Brain Stimulation (Placebo) (Sham Comparator): Participants will receive sham stimulation (placebo) using high-definition tDCS
  Interventions: Device: transcranial direct-current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct-current stimulation (tDCS) — 20 minutes duration using high-definition system with center-surround configuration
  Other Names: Transcranial electrical stimulation

SUMMARY:
This study will determine whether transcranial direct current stimulation (tDCS) can be used alter the amplitude of spontaneous neural activity, and thereby modulate cognitive function in healthy adults

DETAILED DESCRIPTION:
An emerging neurological tool, called transcranial Direct Current Stimulation (tDCS), has recently been shown to safely and effectively enhance cognition in healthy individuals, as well as reduce key symptomatology in disorders such as stroke and depression, with only negligible side effects. tDCS delivers low-amplitude current to the scalp using small electrodes and part of this current passes through the skull and modulates neural activity in the underlying brain region. How this tiny amount of electric current acts to improve cognitive function and reduce symptoms (e.g., motor impairments in stroke patients with a lesion in motor brain areas) is currently unknown, although many investigators across the world are now working on this problem. Magnetoencephalography (MEG) offers a unique view of neural function, as it can delineate changes in active brain regions with excellent temporal resolution (< 1 ms) and high spatial accuracy (2-3 mm). MEG non-invasively measures the magnetic fields that emanate from active neocortical cells. The potential of the MEG technique to precisely monitor the neural effects of tDCS shows extreme promise, but to date the method has been rarely utilized in this area.

Under this protocol, Modulation of Spontaneous Cortical Activity by tDCS: BRAIN Initiative I, approximately 124 participants will provide written informed consent, undergo cognitive and behavioral testing and a structural MRI during a single visit, and then return several weeks later (2-4 weeks) to complete a short tDCS session followed by a MEG recording (i.e., after tDCS). Most participants will return for two more visits, each separated by 2-4 weeks, that include a tDCS session followed by a MEG recording (i.e., 4 total visits). The three tDCS-MEG visits will be identical except that the nature of the stimulation (e.g., location, amplitude, direction/polarity) will be different.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the participant.
* Age: 19-35 years of age at enrollment or 55-72 years of age at enrollment.
* Gender: males and females included.
* Right-handed based on the Edinburgh Handedness Inventory
* Cognitive functioning: Intelligent Quotient (IQ) of 85 - 115 on the Wechsler Adult Intelligence Scale-Revised
* Ability to complete the questionnaires in English, as not all the neuropsychological tests and questionnaires have been validated in other languages.

Exclusion Criteria:

* Current use of the following medications: psychotropic medications or other medications with significant CNS effects (e.g., antipsychotics, psychostimulants, anticonvulsants, alpha-agonists, adrenergic blockers, lithium, and sedating antihistamines), or other excluded medication.
* Current psychiatric diagnosis based on the Mini-International Neuropsychiatric Interview (MINI) and/or the adult attention-deficit/hyperactivity disorder (ADHD) diagnostic interview.
* Current substance abuse or substance dependence at any time.
* The presence of a known neurological disorder or any major medical illness or injury impacting neurological/psychiatric function (e.g., diabetes, epilepsy, cerebral palsy, traumatic brain injury, significant environmental/toxic injury, neurodegenerative disorder, past meningitis/encephalitis).
* General medical conditions: any major medical conditions that would interfere with involvement in the study or may affect central nervous system (CNS) function as judged by the investigative team.
* History of clinically-significant head trauma.
* Pregnancy
* Any other condition that, in the opinion of the investigator, is a contraindication to participation
* The presence of any ferrous metal implant, including orthodontics (e.g., braces), which may interfere with the MEG data acquisition and/or be a MRI safety concern.
* Inability to correct visual acuity to 20/20 with corrective lenses (we can correct from +5 to -6 diopters in .5 diopter steps, separately for each eye, with non-magnetic corrective lenses in the laboratory).

Ages: 19 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony W Wilson, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, de-identified data from this study will be stored in the National Institute of Mental Health's (NIMH) Data Archive.
Supporting Information: Study Protocol
Time Frame: Data will be fully updated by the end of the study and will remain publicly available indefinitely.
Access Criteria: Approval/Account from the NIMH

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that 133 participants were enrolled using a cross-over design and randomized into one of six tracks. There was at least a 7 day washout between each of the three visits and this was the same across the six tracks.
Groups:
- Anodal Stimulation, Then Cathodal Stimulation, Then Sham: Participants received 20 minutes of anodal stimulation using high-definition transcranial direct-current stimulation (HD-tDCS). At least seven days later, they received 20 minutes of cathodal stimulation using HD-tDCS. At least seven days later, they received 20 minutes of sham stimulation using HD-tDCS.
- Anodal Stimulation, Then Sham Stimulation, Then Cathodal Stimulation: Participants received 20 minutes of anodal stimulation using high-definition transcranial direct-current stimulation (HD-tDCS). At least seven days later, they received 20 minutes of sham stimulation using HD-tDCS. At least seven days later, they received 20 minutes of cathodal stimulation using HD-tDCS.
- Cathodal Stimulation, Then Anodal Stimulation, Then Sham: Participants received 20 minutes of cathodal stimulation using high-definition transcranial direct-current stimulation (HD-tDCS). At least seven days later, they received 20 minutes of anodal stimulation using HD-tDCS. At least seven days later, they received 20 minutes of sham stimulation using HD-tDCS.
- Cathodal Stimulation, Then Sham, Then Anodal Stimulation: Participants received 20 minutes of cathodal stimulation using high-definition transcranial direct-current stimulation (HD-tDCS). At least seven days later, they received 20 minutes of sham stimulation using HD-tDCS. At least seven days later, they received 20 minutes of anodal stimulation using HD-tDCS.
- Sham Stimulation, Then Anodal Stimulation, Then Cathodal Stimulation: Participants received 20 minutes of sham stimulation using high-definition transcranial direct-current stimulation (HD-tDCS). At least seven days later, they received 20 minutes of anodal stimulation using HD-tDCS. At least seven days later, they received 20 minutes of cathodal stimulation using HD-tDCS.
- Sham Stimulation, Then Cathodal Stimulation, Then Anodal Stimulation: Participants received 20 minutes of sham stimulation using high-definition transcranial direct-current stimulation (HD-tDCS). At least seven days later, they received 20 minutes of cathodal stimulation using HD-tDCS. At least seven days later, they received 20 minutes of anodal stimulation using HD-tDCS.
Period: Overall Study
Arm/Group | Anodal Stimulation, Then Cathodal Stimulation, Then Sham | Anodal Stimulation, Then Sham Stimulation, Then Cathodal Stimulation | Cathodal Stimulation, Then Anodal Stimulation, Then Sham | Cathodal Stimulation, Then Sham, Then Anodal Stimulation | Sham Stimulation, Then Anodal Stimulation, Then Cathodal Stimulation | Sham Stimulation, Then Cathodal Stimulation, Then Anodal Stimulation
Started | 22 | 22 | 22 | 23 | 22 | 22
Completed | 21 | 21 | 20 | 21 | 20 | 21
Not Completed | 1 | 1 | 2 | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Of the 133 enrolled, 124 participants completed all interventions. The order of interventions was balanced and the goal was to identify the impact of the intervention and eliminate any effect of administration order.
Groups:
- All Study Participants: All participants received all interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] — Age at enrollment in years; self-reported
  years | 44 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 110
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 101
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 124
Mental health questionnaire [Count of Participants; unit: Participants] — This was a 20 item pass/fail screener for psychiatric disease and cognitive impairment; participants had to pass screen ruling out psychiatric disease and cognitive impairment to be included in the study. If they endorsed being previously diagnosed with any psychiatric or neurological condition, including substance use disorders, they were excluded from the study. In total, 133 participants passed the screener and started the full study. However, only 124 completed all study aspects and participants had to complete all aspects to be included in the final analyses.
  Participants | 124

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Performance (Accuracy) on Cognitive Tests of Perceptual Processing
Description: Do participants perform better in terms of accuracy following tDCS on behavioral measures of perceptual processing.
Time Frame: During the 90 minutes following stimulation
Population: 124 participants completed all three conditions (anodal, cathodal, sham) and have evaluable data.
Measure: Mean (Standard Deviation); unit: percent correct
Groups:
- Anodal Stimulation: Participants will receive 20 minutes of anodal stimulation using high-definition transcranial direct-current stimulation (tDCS) with center-surround configuration
- Cathodal Stimulation: Participants will receive 20 minutes of cathodal stimulation using high-definition transcranial direct-current stimulation (tDCS) with center-surround configuration
- Sham Stimulation (Placebo): Participants will receive 20 minutes of sham stimulation using high-definition transcranial direct-current stimulation (tDCS) with center-surround configuration
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham Stimulation (Placebo)
Number analyzed (Participants) | 124 | 124 | 124
percent correct | 97 (1.26) | 98 (1.05) | 98 (.94)

2. Secondary Outcome: The Power of Spontaneous Alpha Activity as Quantified by MEG Imaging
Description: Does spontaneous alpha (9-13 Hz) power, as measured by MEG, get stronger following tDCS. Spontaneous activity refers to the level of background neural activity and is typically divided into frequency bands (e.g., alpha, gamma) that reflect the number of cycles per second. The outcome measure unit is nano-amperes square (nA^2) since source-resolved MEG measures reflect electric current strength and not voltage units as in electroencephalography (EEG). The square is necessary since we examined power, which is the square of amplitude in the frequency domain. The unit is also commonly expressed as nAm^2 since the strength of the electric current is over a defined length.
Time Frame: During the 90 minutes following stimulation
Population: 124 participants completed all three conditions (anodal, cathodal, sham) and have evaluable data.
Measure: Mean (Standard Error); unit: nano-amperes square (nA^2)
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham Stimulation (Placebo)
Number analyzed (Participants) | 124 | 124 | 124
nano-amperes square (nA^2) | 23.26 (3.06) | 15.88 (2.18) | 17.02 (2.46)

3. Secondary Outcome: The Power of Oscillatory Alpha Activity as Quantified by MEG Imaging
Description: Does oscillatory alpha neural activity, as measured by MEG, get stronger following tDCS. Oscillatory activity refers band-limited increases or decreases in the power of neural activity, relative to baseline, in response to a stimulus.
Time Frame: During the 90 minutes following stimulation
Population: 124 participants completed all three conditions (anodal, cathodal, sham) and have evaluable data.
Measure: Mean (Standard Error); unit: percent increase/decrease from baseline
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham Stimulation (Placebo)
Number analyzed (Participants) | 124 | 124 | 124
percent increase/decrease from baseline | -27.34 (3.18) | -26.10 (3.03) | -30.88 (5.11)

4. Primary Outcome: Behavioral Performance (Reaction Time) on Cognitive Tests of Perceptual Processing
Description: Do participants perform better in terms of reaction time following tDCS on behavioral measures of perceptual processing.
Time Frame: During the 90 minutes following stimulation
Population: 124 participants completed all three conditions (anodal, cathodal, sham) and have evaluable data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham Stimulation (Placebo)
Number analyzed (Participants) | 124 | 124 | 124
milliseconds | 713 (67) | 708 (58) | 724 (52)

5. Secondary Outcome: The Power of Spontaneous Gamma Activity as Quantified by MEG Imaging
Description: Does spontaneous gamma (45-80 Hz) power, as measured by MEG, get stronger following tDCS. Spontaneous activity refers to the level of background neural activity and is typically divided into frequency bands (e.g., alpha, gamma) that reflect the number of cycles per second. The outcome measure unit is nano-amperes square (nA^2) since source-resolved MEG measures reflect electric current strength and not voltage units as in electroencephalography (EEG). The square is necessary since we examined power, which is the square of amplitude in the frequency domain. The unit is also commonly expressed as nAm^2 since the strength of the electric current is over a defined length.
Time Frame: During the 90 minutes following stimulation
Population: 124 participants completed all three conditions (anodal, cathodal, sham) and have evaluable data.
Measure: Mean (Standard Error); unit: nano-amperes square (nA^2)
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham Stimulation (Placebo)
Number analyzed (Participants) | 124 | 124 | 124
nano-amperes square (nA^2) | 3.46 (1.74) | 3.30 (1.89) | 2.43 (1.55)

6. Secondary Outcome: The Power of Oscillatory Gamma Activity as Quantified by MEG Imaging
Description: Does oscillatory gamma neural activity, as measured by MEG, get stronger following tDCS. Oscillatory activity refers band-limited increases or decreases in the power of neural activity, relative to baseline, in response to a stimulus.
Time Frame: During the 90 minutes following stimulation
Population: 124 participants completed all three conditions (anodal, cathodal, sham) and have evaluable data.
Measure: Mean (Standard Error); unit: percent increase/decrease from baseline
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham Stimulation (Placebo)
Number analyzed (Participants) | 124 | 124 | 124
percent increase/decrease from baseline | 10.78 (2.74) | 6.35 (1.98) | 6.28 (1.87)

ADVERSE EVENTS:
Time Frame: Each participant was in the study for about one month (4 weeks).
Description: Standard definitions for adverse events were used.
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham Stimulation (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/133 | 0/133
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/133 | 0/133
Other Adverse Events (participants affected / at risk) | 0/133 | 0/133 | 0/133

LIMITATIONS AND CAVEATS:
Focus on single stimulation amplitude and duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT03672747/Prot_SAP_001.pdf